CLINICAL TRIAL: NCT06102642
Title: The Clinical Usage of a Free Gingival Graft Combined With Frenotomy in Patients With High Frenal Attachment: A Clinical Case Series
Brief Title: The Clinical Usage of a Free Gingival Graft Combined With Frenotomy in Patients With High Frenal Attachment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Saleh Saleh Saleh, Master degree student, periodontology department, faculty of dentistry, Cairo University., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MohSaleh123
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: High Frenum Attachment; Free Gingival Graft
Keywords: Frenotomy; Free gingival graft; High frenum attachment; Frenal relocation

STUDY DESIGN:
Intervention Model Description: Case Series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combining Free Gingival Graft with frenotomy procedure (Experimental): evaluate the usage of free gingival graft combined with frenotomy in order to measure the gain in the width of keratinized gingiva, relapse, mucosal healing and postoperative pain.
  Interventions: Biological: Combining free gingival graft with frenotomy procedure

INTERVENTIONS:
Biological: Combining free gingival graft with frenotomy procedure — The aim of the study is to evaluate the usage of free gingival graft combined with frenotomy in order to measure the gain in the width of keratinized gingiva, relapse, mucosal healing and postoperative pain.

SUMMARY:
In patients with high frenal attachment will placement of free gingival graft combined with frenotomy result in gain of width of keratinized gingiva, decrease relapse, improve mucosal healing and have acceptable postoperative pain?

DETAILED DESCRIPTION:
In patients with high frenal attachment will placement of free gingival graft combined with frenotomy result in gain of width of keratinized gingiva, decrease relapse, improve mucosal healing and have acceptable postoperative pain?

To the best of our knowledge there aren't any studies discussing the use of free gingival graft in combination with frenotomy procedure to decrease relapse & morbidity of the condition; thus the objective of this case series study is to evaluate the effectiveness of using free gingival graft in combination with frenotomy procedure on increasing the width of keratinized tissue & decreasing relapse, postoperative pain and scar formation.

Inclusion criteria:

Ages 18-40 years old Systemically healthy Gingival and plaque index <10 Good oral hygiene Highly attached mandibular labial frenum. Narrow sulcus depth Thin gingival phenotype

Exclusion criteria:

Smokers Poor oral hygiene Patient with a physical disability that hinders the upkeep of good oral hygiene measures.

Taking any medications that could affect healing Any systemic diseases that delay wound healing. Deep sulcus Thick gingival phenotype Pervious frenal procedures Pregnant or lactating females Pervious periodontal surgery within the last 6 months before the start of the trial

Interventions

Preoperative measures:

1. All subjects will pass through phase I therapy (Supragingival scaling, subgingival debridement and oral hygiene instructions) before any surgical procedures.
2. After 4 weeks, all subjects will be examined to determine patient compliance with oral hygiene procedures (tooth brushing twice daily and chlorhexidine HCL 1.25% mouthwash twice daily).
3. Eligible & complied patients will be enrolled in the study

Intervention - Surgical Phase (T0):

1. The same operator (M S) will perform all procedures.
2. After following complete aseptic precautions, surgical technique will be performed. Local infiltration will be done using local anaesthetic solution 4% articaine with 1/200 000 adrenaline solution.
3. A horizontal incision will be placed at mucogingival junction using 15c blade with respect to teeth 42,41,31,32, which is then followed by supraperiosteal dissection or frenal relocation of the mandibular labial frenum up to the desired level using periosteal elevator.
4. Undermining the edges of the frenum using periosteal elevator separating the epithelium from the underlining lip mucosa.
5. The mucosa is sutured in the periosteum by using simple interrupted suture at the desired new level of the frenum.
6. Gauze moistened with saline is to be placed over the recipient bed until graft placement.
7. A free gingival autograft will be harvested from the palate using 15c blade and tissue forceps.
8. Stabilization of the free gingival autograft in place using a 6-0 resorbable Vicryl suture using combination of interrupted and sling sutures.

Post-operative care:

1. Patients abstained from tooth brushing for 2 days post-operatively.
2. Using 0.2% cholohexidine mouthwash twice daily for 14 days to be started on the 2nd day of surgery.
3. Ibuprofen 600 mg 1 tablet PRN.
4. Patients will be instructed to:

   1. Follow the instructions completely.
   2. Keep up a strict follow-up schedule.
   3. Brush their teeth twice a day, with a soft brush, and avoid brushing the surgical area (to be started 2 days post-surgery).
   4. Not to touch the surgical area, with the tongue or fingers.
   5. Do not wear any kind of dental appliances, on or around the surgical site.
   6. Not to eat or bite on the anterior teeth during the healing period.

Follow-up (T1, T2,T3, T4):

T1 1. Patients recalled after 5 days for measurement of mucosal healing using IPR (Inflammatory, Proliferativ, & Remodeling) Wound Healing Scale (Hamzani & Chaushu, 2018).

T2

1. Patients recalled after 14 days for suture removal.
2. Measurement of pain score using Numerical Rating scale (NRS) measurement. (Williamson & Hoggart, 2005).
3. Measurement of mucosal healing using IPR (Inflammatory, Proliferativ, & Remodeling) Wound Healing Scale (Hamzani & Chaushu, 2018).

T3

1. Patients recalled after 2 months.
2. Measurement of mucosal healing using IPR (Inflammatory, Proliferativ, & Remodeling) Wound Healing Scale (Hamzani & Chaushu, 2018).

T4

1. Patients recalled after 3 months for the evaluation of frenum relapse using periodontal probe (Sarmadi et al., 2021).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-40 years old
* Systemically healthy
* Gingival and plaque index <10
* Good oral hygiene
* Highly attached mandibular labial frenum.
* Narrow sulcus depth
* Thin gingival phenotype

Exclusion Criteria:

* Smokers
* Poor oral hygiene
* Patient with a physical disability that hinders the upkeep of good oral hygiene measures.
* Taking any medications that could affect healing
* Any systemic diseases that delay wound healing.
* Deep sulcus
* Thick gingival phenotype
* Pervious frenal procedures
* Pregnant or lactating females
* Pervious periodontal surgery within the last 6 months before the start of the trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Width of keratinized tissue | T1: 5days post-surgery, T2:14 days post-surgery, T3: 2months post-surgery & T4: 3months post-surgery.
  It will be measured using periodontal probe at T1, T2, T3 and T4

SECONDARY OUTCOMES:
Mucosal healing | T1: 5days post-surgery, T2:14 days post-surgery, T3: 2months post-surgery
  it will be measured using IPR (Inflammatory Proliferative Remodeling) Wound Healing Scale at T1, T2 and T3.
Post-operative pain | T2:14 days post-surgery.
  it will be measured using Numerical Rating scale (NRS) at T2
Relapse | T4: 3months post-surgery.
  it will be measured using periodontal probe at T4

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Cairo University; Nada Zazou, Ass Lecturer, Study Chair — MSA University